CLINICAL TRIAL: NCT06249165
Title: VictORION-INCLUSION: Evaluating INClisiran as a soLUtion to Improve LDL-C Management and cloSe Care Gaps in an Inclusive ASCVD and ASCVD Risk Equivalent populatiON
Brief Title: VictORION-INCLUSION: Evaluating Inclisiran for Cholesterol Managment in Heart Disease
Acronym: V-INCLUSION
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115658; CKJX839A1US10 (Other: Novartis)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Hyperlipidemia; Secondary Cardiovascular Prevention; Primary Prevention; Atherosclerotic Cardiovascular Disease (ASCVD); Hypercholesterolemia; Lipid lowering therapies; Inclisiran
MeSH Terms: conditions — Atherosclerosis; Hyperlipidemias; Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Intervention Model Description: randomized, controlled, multicenter, open-label two arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Inclisiran (Experimental): Inclisiran + Usual Care
  Interventions: Drug: Inclisiran
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Drug: Inclisiran — Inclisiran sodium 300 mg/1.5 ml (equivalent to 284 mg inclisiran liquid) in prefilled syringe (PFS).
  Other Names: Leqvio
  Arms: Inclisiran

SUMMARY:
VictORION-INCLUSION (V-INCLUSION) seeks to evaluate the effectiveness of inclisiran as an innovative therapy with the potential to help bridge care gaps in historically understudied and undertreated populations by leveraging electronic health records (EHR) in multiple US Healthcare Systems (HCS) to systematically identify those at high risk for and already diagnosed with ASCVD for more expeditious achievement of LDL-C targets.

DETAILED DESCRIPTION:
The trial consists of two parts. Part 1 is a randomized, controlled, multicenter, open-label two arm trial comparing inclisiran and usual care versus usual care alone in an inclusive study population identified by electronic health records. Part 2 is a single arm trial consisting of Part 1 usual care participants initiating inclisiran at Day 360, and receiving two additional doses on day 450 and 630 (dosed in similar fashion to inclisiran + UC arm in Part 1). Approximately 1440 participants will be randomized to either inclisiran + usual care or to usual care only. Eligible participants must be at high risk for or be diagnosed with established ASCVD (prior CAD, PAD, CeVD event) and LDL-C above treatment threshold despite treatment with statin therapy (or with documented statin intolerance).

The study funder made a business decision to close the study to enrollment. Any patients identified and confirmed eligible prior to May 30, 2025 were permitted to be randomized through June 6, 2025. A total of 130 participants were enrolled. Participants randomized to Inclisiran + Usual Care will complete the study as originally planned. Participants randomized to Usual Care alone will have the option to receive inclisiran earlier if they choose to do so. They may also opt to complete only the Usual Care portion of the study (i.e., never receive study inclisiran) or to withdraw from the study. Usual Care participants will be required to sign an addendum to consent to these changes and identify their selection.

The study population will consist of underrepresented and historically understudied male and female participants (targeting 50% female, 70% underrepresented [Black/African American, Hispanic/Latino, Asian, other] and 10% rural participants of any sex or race/ethnicity) ≥18 years of age with a history of ASCVD (coronary artery disease, ischemic cerebrovascular disease or peripheral arterial disease) or ASCVD risk equivalent (HeFH, Type 2 DM, or 10 year ASCVD risk score ≥ 20%) who have elevated LDL-C (≥ 70 mg/dL or LDL-C ≥ 100 mg/dL) respectively) despite being treated with statin therapy. A total of approximately 1440 participants will be randomized to inclisiran + usual care or usual care in a 1:1 ratio at up to 30 US healthcare systems.

ELIGIBILITY:
Inclusion Criteria: Must meet all criteria below.

1. Males and females >= 18 years of age
2. Have clinical ASCVD or ASCVD risk equivalent diagnosis captured in EHR
3. Serum LDL-C ≥ 70 mg/dL for participants with ASCVD, or LDL-C ≥ 100 mg/dL for ASCVD risk equivalent participants, based on last recorded LDL-C value within the preceding eighteen (18) months without a subsequent change in lipid lowering therapy.
4. Willing and able to give informed consent before initiation of any study related procedures and willing to comply with all required study procedures.
5. On statin therapy, or have documented statin intolerance, as determined by the treating clinician. Participants for whom statin therapy has been recently initiated must be on stable therapy for at least 4 weeks and subsequent LDL-C must be above the threshold.
6. From historically underrepresented populations in cardiovascular clinical research, including at least one of the following: female sex; Hispanic/Latino ethnicity; Black/African-American, Asian, or Native American race; rural dwelling based on the HRSA definition for determining rural grant eligibility using the Federal Office of Rural Health Policy (FORHP) 2010 County and Census Tract file.

Exclusion Criteria: Cannot meet any criteria below.

1. Planned use of other investigational products or devices during the course of the study.
2. Treatment with monoclonal antibodies directed towards PCSK9 within 90 days or with inclisiran within 180 days of pre-screening.
3. History of hypersensitivity to the study treatment or its excipients or to other siRNA drugs.
4. Pregnant or nursing (lactating) women.
5. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment.
6. New York Heart Association (NYHA) class III or IV heart failure or last known left ventricular ejection fraction <25%.
7. Significant cardiac arrhythmia within 3 months prior to randomization that is not controlled by medication or other methods (i.e. via ablation etc.) at the time of pre-screening. Controlled arrhythmia is not an exclusion.
8. Uncontrolled hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to randomization despite antihypertensive therapy.
9. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or alanine aminotransferase (ALT) elevation >3x ULN, aspartate aminotransferase (AST) elevation >3x ULN, or total bilirubin elevation >2x ULN (except participants with Gilbert's syndrome) at pre-screening confirmed by a repeat measurement at least one week apart. Lack of repeat measurement is not considered an exclusion.
10. End-stage renal disease (ESRD), defined as being on dialysis of any kind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Achievement of LDL-C targets | Day 360
  Achieving LDL-C targets (LDL-C < 70 mg/dL for ASCVD participants or LDL-C < 100 for ASCVD risk equivalent participants) (yes/no)

SECONDARY OUTCOMES:
Achievement of LDL-C targets by subgroup | Day 360
  Achieving LDL-C targets at Day 360 in the following participant subgroups: Female, Black/African American, Hispanic/Latino, Rural.
Change in LDL-C from baseline by population | Day 360
  Change in LDL-C value from baseline (absolute change, percent change, average absolute change, average percent change) in entire population, ASCVD population, and ASCVD risk equivalent population
Achievement of LDL-C targets by population | Day 360
  Achieving LDL-C target at day 360 in ASCVD population and ASCVD risk equivalent population
Safety and tolerability of inclisiran | Through study completion, up to approximately 630 days
  Incidence of AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Neha Pagidipati, MD, Principal Investigator — Duke Clinical Research Institute
Locations (23):
- United States (23):
  - Univ. of Alabama - Birmingham, Birmingham, Alabama
  - Univ. of California - Irvine, Orange, California
  - San Francisco General Hospital, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Wellstar Paulding, Hiram, Georgia
  - Rush University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - JHU - Suburban Hospital, Bethesda, Maryland
  - Johns Hopkins, Columbia, Maryland
  - Essentia Health, Duluth, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Heart House of NJ, Haddon Heights, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Medical Univ. of South Carolina, Charleston, South Carolina
  - Houston Methodist, Houston, Texas
  - Baylor Scott & White - Waco, Waco, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No